CLINICAL TRIAL: NCT01556282
Title: A Humanitarian Device Exemption Treatment Protocol of TheraSphere for Treatment of Unresectable Hepatocellular Carcinoma in Patients With Portal Vein Thrombosis
Brief Title: TheraSpheres Treatment for Unresectable Hepatocarcinoma and Portal Vein Thrombosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Hyun Kevin Kim, MD,FSIR Director of Interventional Radiology and Image Guided Medicine, Emory University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00015167
Record Dates: First submitted 2012-02-13; First posted 2012-03-16 (Estimated); Last update posted 2014-05-28 (Estimated); Status verified 2014-05

CONDITIONS: Liver Cancer; Portal Vein Thrombosis
Keywords: Hepatocellular Carcinoma; portal vein thrombosis; HCC
MeSH Terms: conditions — Liver Neoplasms; Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Therasphere (Experimental)
  Interventions: Device: TheraSphere

INTERVENTIONS:
Device: TheraSphere — TheraSphere are microspheres with y-90 a radioactive material that will be injected into the liver through a blood vessel.
  Other Names: There are no other names for this device.

SUMMARY:
Therasphere will be administered via catheter through the Hepatic Artery to treat patients with Hepatocellular Carcinoma and Portal vein Thrombosis.

DETAILED DESCRIPTION:
Therasphere consists of glass microspheres containing a radioactive material called Yttrium-90.

Therasphere is delivered into the liver tumor through a catheter placed into the hepatic artery which is the artery that provides the main blood supply to the tumor, this way delivering the radioactive material directly to the tumor and sparing the rest of the liver tissue from radiation.

ELIGIBILITY:
Inclusion Criteria:

* 18 yrs of age or older
* Diagnosis of Hepatocellular Carcinoma
* Portal Vein Thrombosis
* ECOG performance < 2

  ->4 weeks since prior radiation, surgery or chemotherapy.
* Life expectancy > 3 months
* Able to provide written informed consent process in accordance with institutional review boards guidelines.

Exclusion Criteria:

* Contraindications to angiography and selective visceral catheterization.
* Evidence of blood flow to the lung from the liver greater than 16.5 mCi
* Evidence of any detectable Tc-99m MAA flow to the stomach or duodenum, after application of established angiographic techniques to stop or mitigate such flow.
* Significant extrahepatic disease.
* Severe liver disfunction of pulmonary insufficiency.
* Active uncontrolled infection.
* Significant underlying medical or psychiatric illness.
* Pregnancy. Patients will be excluded if they have pre-existing diarrhea/illness, or if they have a co-morbid disease or condition that would preclude safe delivery of TheraSphere treatment and place the patient at undue risk.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2009-03; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Response rate to the administration of Therasphere | Participants will be followed through 1 year after the procedure at 1 month, 3 months, 6 months and 1 year visits

SECONDARY OUTCOMES:
Progression free survival for patients with unresectable liver cancer. | Participants will be followed through 1 year after receiving treatment
  Patients will be followed after treatment at 1 month, 3 months, 6 months, and 1 year.

CONTACTS AND LOCATIONS:
Overall Officials: Hyun s Kim, MD, Principal Investigator — Emory University
Locations (1):
- Emory University Hospital, Atlanta, Georgia, United States

REFERENCES:
- [Derived] Xing M, Kokabi N, Camacho JC, Kim HS. Prospective longitudinal quality of life and survival outcomes in patients with advanced infiltrative hepatocellular carcinoma and portal vein thrombosis treated with Yttrium-90 radioembolization. BMC Cancer. 2018 Jan 12;18(1):75. doi: 10.1186/s12885-017-3921-1. PMID 29329568
- [Derived] Kokabi N, Camacho JC, Xing M, El-Rayes BF, Spivey JR, Knechtle SJ, Kim HS. Open-label prospective study of the safety and efficacy of glass-based yttrium 90 radioembolization for infiltrative hepatocellular carcinoma with portal vein thrombosis. Cancer. 2015 Jul 1;121(13):2164-74. doi: 10.1002/cncr.29275. Epub 2015 Apr 6. PMID 25847227